CLINICAL TRIAL: NCT02249000
Title: Safety and Clinical Performance of the Self-expanding Transcatheter BIOVALVE Prosthesis in Subjects With Severe Symptomatic Aortic Stenosis Suitable for Transfemoral Transcatheter Aortic Valve Implantation
Brief Title: BIOVALVE - I / II Clincial Investigation
Acronym: BIOVALVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik AG (Industry)
Collaborators: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1205
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Last update posted 2024-06-11 (Actual); Status verified 2019-01

CONDITIONS: Heart Valve Diseases; Aortic Valve Stenosis
MeSH Terms: conditions — Heart Valve Diseases; Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BIOVALVE prosthesis (Experimental): Transcatheter Aortic Valve Replacement (TAVR)
  Interventions: Device: BIOVALVE prosthesis

INTERVENTIONS:
Device: BIOVALVE prosthesis — Transcatheter Aortic Valve Replacement (TAVR)

SUMMARY:
First-in-Human clinical investigation to evaluate the safety and clinical performance of the BIOVALVE prosthesis in subjects presenting with severe symptomatic aortic valve stenosis, which are as judged by the heart team, indicated for transfemoral transcatheter aortic valve implantation

DETAILED DESCRIPTION:
In a non-randomized, prospective, multi-center clinical investigation, approximately 86 eligible subjects will be enrolled.

Phase 1: BIOVALVE-I feasibility clinical investigation: Approximately 13 eligible subjects will be enrolled.

Phase 2: BIOVALVE-II pilot clinical investigation: Approximately 73 eligible subjects will be enrolled.

BIOVALVE-I/II subjects follow the same clinical investigation plan (CIP) in all aspects.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is ≥65 years
2. The subject has provided written informed consent
3. Subject is willing to participate in the clinical investigation and to comply with all of the study procedures and follow-up visits
4. NHYA class ≥II
5. High surgical risk: Logistic EuroSCORE-I ≥20% (or equivalence of EuroSCORE-II) or STS score ≥10% or co-morbidity judged by the heart team (consisting of at least one interventional cardiologist and one cardiac surgeon) to pose an absolute or relative contraindication for conventional aortic valve replacement according to VARC-2
6. Severe symptomatic calcific aortic valve stenosis characterized by mean aortic gradient >40 mm Hg or peak jet velocity >4.0 m/s or effective orifice area (EOA) of <1.0 cm2 (<0.6 cm2/m2 body surface area)
7. Annulus diameter as determined by multi-slice computed tomography (MSCT) from 23-26 mm

Exclusion Criteria:

1. Trans-esophageal echocardiogram (TEE) is contraindicated
2. Congenital bicuspid or unicuspid valve
3. Left ventricular outflow tract (LVOT) obstruction such as hypertrophic obstructive cardio myopathy (HOCM) or subject presenting with systolic anterior motion (SAM). Evidence of intra cardiac mass, thrombus or vegetation
4. Transfemoral access vessel characteristics that would preclude safe placement of a 18 French sheath
5. Vessel and/or anatomical characteristics that would preclude safe delivery of the BIOVALVE prosthesis to the ascending aorta and/or placement of the prosthesis
6. Anatomical restrictions such as shallow sinuses with heavily calcified leaflets, low height of coronary ostia, extreme tortuosity of the aortic arch, thoracic (TAA) or abdominal (AAA) aortic aneurysm, presence of endovascular stent graft
7. Severe mitral regurgitation grade >3
8. Severe mitral stenosis
9. Prosthetic mitral valve
10. Severe left ventricular dysfunction with left ventricular ejection fraction (LVEF) <20%
11. Hemodynamic instability
12. Percutaneous coronary intervention (PCI) within 30 days prior to index procedure and / or planned PCI during index procedure
13. Renal insufficiency (creatinine >2.5 mg/dl) or subject under dialysis and/or renal replacement therapy
14. Any cerebrovascular event or transient ischemic attack (TIA) within 180 days prior to TAVI procedure
15. Evidence of acute myocardial infarction (defined as ≥2 fold CK level or in absence of CK a ≥3 fold CKMB level above the upper range limit within ≤30 days prior to TAVI procedure)
16. Blood dyscrasia defined as: leucopenia (WBC <1000 mm³), thrombocytopenia (platelet count <50'000 cells/mm³), history of bleeding diathesis requiring blood transfusion
17. Ongoing sepsis or suspected active endocarditis
18. Active peptic ulcer or gastrointestinal bleeding within last 3 months that would preclude anticoagulation
19. Subject refuses blood transfusion
20. Known hypersensitivity to, or contraindication to nitinol, anticoagulation/antiplatelet regimes, any other medications required for the procedure or post-procedure as determined by the heart team, or sensitivity to contrast media which cannot be adequately pre-medicated
21. Need for emergency TAVI intervention, or other medical, social, or psychological conditions that in the opinion of the heart team precludes the subjects from appropriate consent or adherence to protocol required follow-up exams
22. Expectation that subject will not improve despite treatment of aortic stenosis
23. Estimated life expectancy of less than 12 months due to associated non-cardiac co-morbidities
24. Severe pulmonary hypertension (> 60 mm Hg assessed by continuous wave Doppler, TTE) or clinical signs of acute severe right ventricular dysfunction
25. Currently participating in another investigational drug or device study where primary endpoint has not been reached yet

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-09; Primary Completion 2018-03 (Actual); Study Completion 2023-05 (Actual)

PRIMARY OUTCOMES:
Early safety at 30 days (Acc. to VARC-2) | 30 days
  A composite of all-cause mortality, all stroke (disabling/non-disabling), life-threatening bleeding, acute kidney injury stage 2 or 3 (including renal replacement therapy), coronary artery obstruction requiring intervention, major vascular complication and valve-related dysfunction requiring repeat procedure (balloon aortic valvuloplasty (BAV), transcatheter aortic valve implantation (TAVI), or surgical aortic valve replacement (SAVR)).

SECONDARY OUTCOMES:
Combined safety endpoint at 30 days (Acc. to VARC-1) | 30 days
  A composite of all-cause mortality, major stroke, life-threatening (or disabling) bleeding, acute kidney injury stage 3 (including renal replacement therapy), peri-procedural myocardial infarction, major vascular complication and repeat procedure for valve-related dysfunction (surgical or interventional therapy)
Clinical efficacy after 30 days (Acc. to VARC-2): | 30 days
  A composite of all-cause mortality, all stroke (disabling and non-disabling), requiring hospitalizations for valve-related symptoms or worsening congestive heart failure, NYHA class III or IV, valve-related dysfunction (mean aortic valve gradient ≥20 mm Hg, effective orifice area (EOA) ≤0.9-1.1 cm2 * and/or Doppler velocity index (DVI) <0.35 m/s, and/or moderate or severe prosthetic valve regurgitation **).
  * depending on body surface area
  ** refers to VARC-2 definitions
Echocardiograhic (ECHO) parameters | Discharge, 30 days, 6 months, 12 months and annually through 5 years
  Effective orifice area (EOA) and effective orifice area index (EOAI) Mean prosthetic valve gradient Prosthetic valve regurgitation (Acc. to VARC-1 and VARC-2)

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Treede, MD, Study Chair — Universitätsklinikum Halle (Saale), Germany; Ulrich Schaefer, MD, Study Chair — University Heart Center Hamburg, Germany
Locations (13):
- ZNA Middelheim, Antwerp, Belgium
- Germany (10):
  - Städtische Kliniken Neuss - Lukaskrankenhaus, Neuss, North Rhine-Westphalia
  - Segeberger Kliniken, Bad Segeberg, Schleswig-Holstein
  - Vivantes Klinikum, Berlin
  - German Heart Center, Berlin
  - University Heart Center, Cologne
  - Universitätsklinikum Halle (Saale), Halle
  - Asklepios Klinik St. Georg, Hamburg
  - University Heart Center, Hamburg
  - Herzzentrum Leipzig, Leipzig
  - Universitätsmedizin Rostock, Rostock
- Catharina-Ziekenhuis, Eindhoven, Netherlands
- Universitätsspital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kappetein AP, Head SJ, Genereux P, Piazza N, van Mieghem NM, Blackstone EH, Brott TG, Cohen DJ, Cutlip DE, van Es GA, Hahn RT, Kirtane AJ, Krucoff MW, Kodali S, Mack MJ, Mehran R, Rodes-Cabau J, Vranckx P, Webb JG, Windecker S, Serruys PW, Leon MB; Valve Academic Research Consortium-2. Updated standardized endpoint definitions for transcatheter aortic valve implantation: the Valve Academic Research Consortium-2 consensus document. EuroIntervention. 2012 Nov 22;8(7):782-95. doi: 10.4244/EIJV8I7A121. PMID 23022744
- [Background] Leon MB, Piazza N, Nikolsky E, Blackstone EH, Cutlip DE, Kappetein AP, Krucoff MW, Mack M, Mehran R, Miller C, Morel MA, Petersen J, Popma JJ, Takkenberg JJ, Vahanian A, van Es GA, Vranckx P, Webb JG, Windecker S, Serruys PW. Standardized endpoint definitions for Transcatheter Aortic Valve Implantation clinical trials: a consensus report from the Valve Academic Research Consortium. J Am Coll Cardiol. 2011 Jan 18;57(3):253-69. doi: 10.1016/j.jacc.2010.12.005. Epub 2011 Jan 7. PMID 21216553
- [Result] Treede H, Lubos E, Conradi L, Deuschl F, Asch FM, Weissman NJ, Schofer N, Schirmer J, Koschyk D, Blankenberg S, Reichenspurner H, Schaefer U. Thirty-day VARC-2 and performance data of a new self-expanding transcatheter aortic heart valve. EuroIntervention. 2015 Nov;11(7):785-92. doi: 10.4244/EIJY15M05_05. PMID 25983028